CLINICAL TRIAL: NCT02169791
Title: A Phase II Trial of Nonmyeloablative Haploidentical Peripheral Blood Stem Cell Transplantation Followed By Maintenance Therapy With the Novel Oral Proteasome Inhibitor, MLN9708, in Patients With High-risk Hematologic Malignancies
Brief Title: Nonmyeloablative Haploidentical Transplant Followed by MLN9708
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NSH 1074; X16035 (Other: Millennium)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Acute Leukemia; Chronic Leukemia; Myelodysplastic Syndrome; Lymphomas; Multiple Myeloma
Keywords: hematologic malignancies
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Hematologic Neoplasms | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haploidentical Transplant (Experimental): All patients will receive a haploidentical donor transplant using a conditioning regimen of Fludarabine (Flu), cyclophosphamide (cy) and total body irradiation (TBI) followed by MLN9708.
  Interventions: Drug: MLN9708

INTERVENTIONS:
Drug: MLN9708 — MLN9708 will be given weekly x 3 weeks every 28 day cycles, for up to 12 cycles starting at D+5 post-transplant.

SUMMARY:
In an attempt to reduce relapse risk and improve outcomes following haploidentical transplantation for patients with high risk hematologic malignancies, the investigators will implement several strategies to augment the well documented effect of NK cell alloreactivity seen in HLA-mismatched transplantation. These strategies include (1) choosing potential haploidentical donors for optimal NK-alloreactivity, (2) utilizing proteasome inhibition post-transplant with MLN9708 to both sensitize tumor cells to NK cytotoxicity and protect against graft-versus-host disease (GVHD), and (3) eliminating mycophenolate mofetil from the post-transplant immunosuppression regimen to improve NK cell reconstitution following haploidentical peripheral blood stem cell transplantation.

DETAILED DESCRIPTION:
Overview of Study Design:

In an attempt to reduce relapse risk and improve outcomes following haploidentical transplantation for patients with high risk hematologic malignancies, the investigators will implement several strategies to augment the well documented effect of NK cell alloreactivity seen in HLA-mismatched transplantation. These strategies include (1) choosing potential haploidentical donors for optimal NK-alloreactivity, (2) utilizing proteasome inhibition post-transplant with MLN9708 to both sensitize tumor cells to NK cytotoxicity and protect against graft-versus-host disease (GVHD), and (3) eliminating mycophenolate mofetil from the post-transplant immunosuppression regimen to improve NK cell reconstitution following haploidentical peripheral blood stem cell transplantation.

Patients will receive a nonmyeloablative haploidentical transplant using a T-cell replete allograft and post-transplant cyclophosphamide as previously described at our center (Bashey et al. J Clin Oncol. 2013; 31(10):1310-6). MLN9708 will be administered once weekly for 3 weeks on a 28 day cycle for one-year post-transplant. Post-transplant immunosuppression will consist of tacrolimus only (MLN9708 will substitute for mycophenolate mofetil as the second GVHD prophylactic medication).

The primary endpoint of this trial will be the risk of relapse and/or progression at one-year post-transplant. Experience from the literature suggests that following a nonmyeloablative haploidentical transplant using post-transplant cyclophosphamide (haplo-pCy), the risk of relapse is approximately 50% at one year post-transplant. It is hoped that under this protocol, this rate will be at most 25%. Thus the investigators statistically formalize this study by testing the null hypothesis that p, the PFS rate is 0.25 or less versus the alternative hypothesis that p is greater than 0.5. A sample size of 25 patients gives 90% power with an alpha=0.05, using the formula for a one sample binomial (two-sided) test of a proportion.

ELIGIBILITY:
Inclusion Criteria:

* Availability of a 3/6 - 5/6 matched (HLA-A, B, DR) related donor
* Donor must have negative HLA cross-match in the host vs. graft direction.
* Donor must be willing to donate mobilized peripheral blood stem cells
* Age ≥ 18 years
* Karnofsky status ≥ 70%
* One of the following high-risk malignancies:
* Chronic Myelogenous Leukemia (chronic phase, resistant and/or intolerant to tyrosine kinase inhibitors (OR) accelerated phase (OR) blast crisis in 2nd chronic phase following induction chemotherapy)
* Acute Myelogenous Leukemia (2nd or subsequent complete remission [CR] (OR) Primary induction chemotherapy failure, but subsequently entered into a CR(OR) 1st CR with poor risk cytogenetics or molecular markers; or arising from preceding hematological disease)
* Myelodysplastic Syndrome (treatment-related, monosomy 7 or complex cytogenetics, IPSS score of 1.5 or greater, Chronic myelomonocytic leukemia [CMML])
* Acute lymphocytic leukemia/lymphoblastic lymphoma (2nd or subsequent CR (OR) Primary induction chemotherapy failure, but subsequently entered into a CR (OR) 1st CR with poor risk cytogenetics)
* Chronic Lymphocytic Leukemia / Prolymphocytic Leukemia (Duration of remission <12 months after receiving chemotherapy with a nucleoside analog (OR) High risk features (i.e. 17p deletion), (OR) Second or subsequent relapse)
* Hodgkin's or Non-Hodgkin's Lymphoma (including low-grade, mantle cell, and intermediate-grade/diffuse) (Previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy or autologous transplantation (AND) Chemoresponsive to most recent salvage therapy
* Multiple Myeloma (Presence of a poor risk cytogenetic abnormality [i.e. 17p, t(4;14)], Relapse post autologous transplant)

Exclusion Criteria:

* Poor cardiac function: left ventricular ejection fraction <40%
* Poor pulmonary function: FEV1, FVC, or DLCO <50% predicted
* Poor liver function: bilirubin >2.5 mg/dl (not due to hemolysis, Gilbert's or primary malignancy), AST/ALT > 3X ULN
* Poor renal function: Creatinine >2.0 mg/dl or creatinine clearance (calculated creatinine clearance is permitted) < 40 mL/min
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* Patients who have any debilitating medical or psychiatric illness which would preclude their giving informed consent or their receiving optimal treatment and follow-up.
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Patient has >/= Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21days of the start of this trial and throughout the duration of this trial.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Szydlo R, Goldman JM, Klein JP, Gale RP, Ash RC, Bach FH, Bradley BA, Casper JT, Flomenberg N, Gajewski JL, Gluckman E, Henslee-Downey PJ, Hows JM, Jacobsen N, Kolb HJ, Lowenberg B, Masaoka T, Rowlings PA, Sondel PM, van Bekkum DW, van Rood JJ, Vowels MR, Zhang MJ, Horowitz MM. Results of allogeneic bone marrow transplants for leukemia using donors other than HLA-identical siblings. J Clin Oncol. 1997 May;15(5):1767-77. doi: 10.1200/JCO.1997.15.5.1767. PMID 9164184
- [Background] Anasetti C, Amos D, Beatty PG, Appelbaum FR, Bensinger W, Buckner CD, Clift R, Doney K, Martin PJ, Mickelson E, et al. Effect of HLA compatibility on engraftment of bone marrow transplants in patients with leukemia or lymphoma. N Engl J Med. 1989 Jan 26;320(4):197-204. doi: 10.1056/NEJM198901263200401. PMID 2643045
- [Background] Anasetti C, Beatty PG, Storb R, Martin PJ, Mori M, Sanders JE, Thomas ED, Hansen JA. Effect of HLA incompatibility on graft-versus-host disease, relapse, and survival after marrow transplantation for patients with leukemia or lymphoma. Hum Immunol. 1990 Oct;29(2):79-91. doi: 10.1016/0198-8859(90)90071-v. PMID 2249952
- [Background] Kanda Y, Chiba S, Hirai H, Sakamaki H, Iseki T, Kodera Y, Karasuno T, Okamoto S, Hirabayashi N, Iwato K, Maruta A, Fujimori Y, Furukawa T, Mineishi S, Matsuo K, Hamajima N, Imamura M. Allogeneic hematopoietic stem cell transplantation from family members other than HLA-identical siblings over the last decade (1991-2000). Blood. 2003 Aug 15;102(4):1541-7. doi: 10.1182/blood-2003-02-0430. Epub 2003 Apr 24. PMID 12714500
- [Background] Kernan NA, Flomenberg N, Dupont B, O'Reilly RJ. Graft rejection in recipients of T-cell-depleted HLA-nonidentical marrow transplants for leukemia. Identification of host-derived antidonor allocytotoxic T lymphocytes. Transplantation. 1987 Jun;43(6):842-7. PMID 3296349
- [Background] Kernan NA, Collins NH, Juliano L, Cartagena T, Dupont B, O'Reilly RJ. Clonable T lymphocytes in T cell-depleted bone marrow transplants correlate with development of graft-v-host disease. Blood. 1986 Sep;68(3):770-3. PMID 3527302
- [Background] Aversa F, Tabilio A, Velardi A, Cunningham I, Terenzi A, Falzetti F, Ruggeri L, Barbabietola G, Aristei C, Latini P, Reisner Y, Martelli MF. Treatment of high-risk acute leukemia with T-cell-depleted stem cells from related donors with one fully mismatched HLA haplotype. N Engl J Med. 1998 Oct 22;339(17):1186-93. doi: 10.1056/NEJM199810223391702. PMID 9780338
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Zuckerman T, Rowe JM. Alternative donor transplantation in acute myeloid leukemia: which source and when? Curr Opin Hematol. 2007 Mar;14(2):152-61. doi: 10.1097/MOH.0b013e328017f64d. PMID 17255793
- [Background] Hallett WH, Ames E, Motarjemi M, Barao I, Shanker A, Tamang DL, Sayers TJ, Hudig D, Murphy WJ. Sensitization of tumor cells to NK cell-mediated killing by proteasome inhibition. J Immunol. 2008 Jan 1;180(1):163-70. doi: 10.4049/jimmunol.180.1.163. PMID 18097016
- [Background] Lundqvist A, Abrams SI, Schrump DS, Alvarez G, Suffredini D, Berg M, Childs R. Bortezomib and depsipeptide sensitize tumors to tumor necrosis factor-related apoptosis-inducing ligand: a novel method to potentiate natural killer cell tumor cytotoxicity. Cancer Res. 2006 Jul 15;66(14):7317-25. doi: 10.1158/0008-5472.CAN-06-0680. PMID 16849582
- [Background] Armeanu S, Krusch M, Baltz KM, Weiss TS, Smirnow I, Steinle A, Lauer UM, Bitzer M, Salih HR. Direct and natural killer cell-mediated antitumor effects of low-dose bortezomib in hepatocellular carcinoma. Clin Cancer Res. 2008 Jun 1;14(11):3520-8. doi: 10.1158/1078-0432.CCR-07-4744. PMID 18519785
- [Background] Sun K, Welniak LA, Panoskaltsis-Mortari A, O'Shaughnessy MJ, Liu H, Barao I, Riordan W, Sitcheran R, Wysocki C, Serody JS, Blazar BR, Sayers TJ, Murphy WJ. Inhibition of acute graft-versus-host disease with retention of graft-versus-tumor effects by the proteasome inhibitor bortezomib. Proc Natl Acad Sci U S A. 2004 May 25;101(21):8120-5. doi: 10.1073/pnas.0401563101. Epub 2004 May 17. PMID 15148407
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Mehta J, Singhal S, Gee AP, Chiang KY, Godder K, Rhee Fv Fv, DeRienzo S, O'Neal W, Lamb L, Henslee-Downey PJ. Bone marrow transplantation from partially HLA-mismatched family donors for acute leukemia: single-center experience of 201 patients. Bone Marrow Transplant. 2004 Feb;33(4):389-96. doi: 10.1038/sj.bmt.1704391. PMID 14716338
- [Background] Lang P, Greil J, Bader P, Handgretinger R, Klingebiel T, Schumm M, Schlegel PG, Feuchtinger T, Pfeiffer M, Scheel-Walter H, Fuhrer M, Martin D, Niethammer D. Long-term outcome after haploidentical stem cell transplantation in children. Blood Cells Mol Dis. 2004 Nov-Dec;33(3):281-7. doi: 10.1016/j.bcmd.2004.08.017. PMID 15528145
- [Background] Waller EK, Giver CR, Rosenthal H, Somani J, Langston AA, Lonial S, Roback JD, Li JM, Hossain MS, Redei I. Facilitating T-cell immune reconstitution after haploidentical transplantation in adults. Blood Cells Mol Dis. 2004 Nov-Dec;33(3):233-7. doi: 10.1016/j.bcmd.2004.08.009. PMID 15528137
- [Background] Guinan EC, Boussiotis VA, Neuberg D, Brennan LL, Hirano N, Nadler LM, Gribben JG. Transplantation of anergic histoincompatible bone marrow allografts. N Engl J Med. 1999 Jun 3;340(22):1704-14. doi: 10.1056/NEJM199906033402202. PMID 10352162
- [Background] Rizzieri DA, Koh LP, Long GD, Gasparetto C, Sullivan KM, Horwitz M, Chute J, Smith C, Gong JZ, Lagoo A, Niedzwiecki D, Dowell JM, Waters-Pick B, Liu C, Marshall D, Vredenburgh JJ, Gockerman J, Decastro C, Moore J, Chao NJ. Partially matched, nonmyeloablative allogeneic transplantation: clinical outcomes and immune reconstitution. J Clin Oncol. 2007 Feb 20;25(6):690-7. doi: 10.1200/JCO.2006.07.0953. Epub 2007 Jan 16. PMID 17228020
- [Background] Fukuda T, Boeckh M, Carter RA, Sandmaier BM, Maris MB, Maloney DG, Martin PJ, Storb RF, Marr KA. Risks and outcomes of invasive fungal infections in recipients of allogeneic hematopoietic stem cell transplants after nonmyeloablative conditioning. Blood. 2003 Aug 1;102(3):827-33. doi: 10.1182/blood-2003-02-0456. Epub 2003 Apr 10. PMID 12689933
- [Background] Dey BR, Spitzer TR. Current status of haploidentical stem cell transplantation. Br J Haematol. 2006 Nov;135(4):423-37. doi: 10.1111/j.1365-2141.2006.06300.x. Epub 2006 Sep 19. PMID 16984391
- [Background] Lehnert S, Rybka WB. Amplification of the graft-versus-host reaction by cyclophosphamide: dependence on timing of drug administration. Bone Marrow Transplant. 1994 Apr;13(4):473-7. PMID 8019473
- [Background] Mayumi H, Umesue M, Nomoto K. Cyclophosphamide-induced immunological tolerance: an overview. Immunobiology. 1996 Jul;195(2):129-39. doi: 10.1016/S0171-2985(96)80033-7. PMID 8877390
- [Background] Mayumi H, Himeno K, Tanaka K, Tokuda N, Fan JL, Nomoto K. Drug-induced tolerance to allografts in mice. XII. The relationships between tolerance, chimerism, and graft-versus-host disease. Transplantation. 1987 Aug;44(2):286-90. doi: 10.1097/00007890-198708000-00021. PMID 3307052
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Lahuerta JJ, Martinez-Lopez J, Serna JD, Blade J, Grande C, Alegre A, Vazquez L, Garcia-Larana J, Sureda A, Rubia JD, Conde E, Martinez R, Perez-Equiza K, Moraleda JM, Leon A, Besalduch J, Cabrera R, Miguel JD, Morales A, Garcia-Ruiz JC, Diaz-Mediavilla J, San-Miguel J. Remission status defined by immunofixation vs. electrophoresis after autologous transplantation has a major impact on the outcome of multiple myeloma patients. Br J Haematol. 2000 May;109(2):438-46. doi: 10.1046/j.1365-2141.2000.02012.x. PMID 10848839
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Kroger N, Zabelina T, Berger J, Duske H, Klyuchnikov E, Binder T, Stubig T, Hilde-brandt Y, Atanackovic D, Alchalby H, Ayuk F, Zander AR, Bacher U, Eiermann T. Donor KIR haplotype B improves progression-free and overall survival after allogeneic hematopoietic stem cell transplantation for multiple myeloma. Leukemia. 2011 Oct;25(10):1657-61. doi: 10.1038/leu.2011.138. Epub 2011 Jun 7. No abstract available. PMID 21647155
- [Background] Shi J, Tricot GJ, Garg TK, Malaviarachchi PA, Szmania SM, Kellum RE, Storrie B, Mulder A, Shaughnessy JD Jr, Barlogie B, van Rhee F. Bortezomib down-regulates the cell-surface expression of HLA class I and enhances natural killer cell-mediated lysis of myeloma. Blood. 2008 Feb 1;111(3):1309-17. doi: 10.1182/blood-2007-03-078535. Epub 2007 Oct 18. PMID 17947507
- [Background] Wu X, Shao Y, Tao Y, Ai G, Wei R, Meng X, Hou J, Han Y, Zhan F, Zheng J, Shi J. Proteasome inhibitor lactacystin augments natural killer cell cytotoxicity of myeloma via downregulation of HLA class I. Biochem Biophys Res Commun. 2011 Nov 11;415(1):187-92. doi: 10.1016/j.bbrc.2011.10.057. Epub 2011 Oct 18. PMID 22033416
- [Background] Ames E, Hallett WH, Murphy WJ. Sensitization of human breast cancer cells to natural killer cell-mediated cytotoxicity by proteasome inhibition. Clin Exp Immunol. 2009 Mar;155(3):504-13. doi: 10.1111/j.1365-2249.2008.03818.x. PMID 19220837
- [Background] Jardine L, Hambleton S, Bigley V, Pagan S, Wang XN, Collin M. Sensitizing primary acute lymphoblastic leukemia to natural killer cell recognition by induction of NKG2D ligands. Leuk Lymphoma. 2013 Jan;54(1):167-73. doi: 10.3109/10428194.2012.708026. Epub 2012 Sep 8. PMID 22742576
- [Background] Vales-Gomez M, Chisholm SE, Cassady-Cain RL, Roda-Navarro P, Reyburn HT. Selective induction of expression of a ligand for the NKG2D receptor by proteasome inhibitors. Cancer Res. 2008 Mar 1;68(5):1546-54. doi: 10.1158/0008-5472.CAN-07-2973. PMID 18316620
- [Background] Blanco B, Perez-Simon JA, Sanchez-Abarca LI, Carvajal-Vergara X, Mateos J, Vidriales B, Lopez-Holgado N, Maiso P, Alberca M, Villaron E, Schenkein D, Pandiella A, San Miguel J. Bortezomib induces selective depletion of alloreactive T lymphocytes and decreases the production of Th1 cytokines. Blood. 2006 May 1;107(9):3575-83. doi: 10.1182/blood-2005-05-2118. Epub 2005 Nov 10. PMID 16282346
- [Background] Blanco B, Perez-Simon JA, Sanchez-Abarca LI, Caballero-Velazquez T, Gutierrez-Cossio S, Hernandez-Campo P, Diez-Campelo M, Herrero-Sanchez C, Rodriguez-Serrano C, Santamaria C, Sanchez-Guijo FM, Del Canizo C, San Miguel JF. Treatment with bortezomib of human CD4+ T cells preserves natural regulatory T cells and allows the emergence of a distinct suppressor T-cell population. Haematologica. 2009 Jul;94(7):975-83. doi: 10.3324/haematol.2008.005017. Epub 2009 Jun 8. PMID 19508976
- [Background] Kim JS, Lee JI, Shin JY, Kim SY, Shin JS, Lim JH, Cho HS, Yoon IH, Kim KH, Kim SJ, Park CG. Bortezomib can suppress activation of rapamycin-resistant memory T cells without affecting regulatory T-cell viability in non-human primates. Transplantation. 2009 Dec 27;88(12):1349-59. doi: 10.1097/TP.0b013e3181bd7b3a. PMID 20029331
- [Background] Blanco B, Sanchez-Abarca LI, Caballero-Velazquez T, Santamaria C, Inoges S, Perez-Simon JA. Depletion of alloreactive T-cells in vitro using the proteasome inhibitor bortezomib preserves the immune response against pathogens. Leuk Res. 2011 Oct;35(10):1412-5. doi: 10.1016/j.leukres.2011.05.018. Epub 2011 Jun 11. PMID 21658766
- [Background] Koreth J, Stevenson KE, Kim HT, McDonough SM, Bindra B, Armand P, Ho VT, Cutler C, Blazar BR, Antin JH, Soiffer RJ, Ritz J, Alyea EP 3rd. Bortezomib-based graft-versus-host disease prophylaxis in HLA-mismatched unrelated donor transplantation. J Clin Oncol. 2012 Sep 10;30(26):3202-8. doi: 10.1200/JCO.2012.42.0984. Epub 2012 Aug 6. PMID 22869883
- [Background] Ohata K, Espinoza JL, Lu X, Kondo Y, Nakao S. Mycophenolic acid inhibits natural killer cell proliferation and cytotoxic function: a possible disadvantage of including mycophenolate mofetil in the graft-versus-host disease prophylaxis regimen. Biol Blood Marrow Transplant. 2011 Feb;17(2):205-13. doi: 10.1016/j.bbmt.2010.08.014. Epub 2010 Aug 22. PMID 20736080
- [Derived] Solomon SR, Solh M, Zhang X, Brown S, Jackson KC, Holland HK, Morris LE, Bashey A. Prospective phase 2 trial of ixazomib after nonmyeloablative haploidentical peripheral blood stem cell transplant. Blood Adv. 2020 Aug 11;4(15):3669-3676. doi: 10.1182/bloodadvances.2020001958. PMID 32777064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was opened at our site 7/15/2014 and closed to accrual on 8/28/18. Patients were recruited internally and were considered if they were undergoing a haploidentical transplant for a high risk malignancy.
Pre-assignment Details: This was a single arm study with no assignment groups. If patients met criteria they were considered for the study. 29 patients were consented and 25 of those patients were deemed eligible to participate. 4 patients were considered screen failures.
Period: Overall Study
Arm/Group | Haploidentical Transplant
Started | 25
Completed (18 patients completed the full study including follow up.) | 18
Not Completed | 7
Not completed — Death | 6
Not completed — patient withdrew consent | 1

BASELINE CHARACTERISTICS:
Population: 25 of those patients were deemed eligible to participate. 4 additional patients were consented but considered screen failures and were not included in the analysis.
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Relapse or Progression
Description: To estimate the incidence of relapse/progression at one-year post-transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
Participants | 10

2. Secondary Outcome: Neutrophil Engraftment
Description: To obtain time to neutrophil engraftment post-transplant
Time Frame: 1 year
Population: All 25 patients were analyzed for time to engraftment
Measure: Median (Full Range); unit: days
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
days | 16 [13 to 27]

3. Secondary Outcome: Time to Platelet Recovery Post Transplant
Description: To measure the time to platelet recovery post-transplant
Time Frame: 1 year
Measure: Median (Full Range); unit: days
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
days | 29 [16 to 47]

4. Secondary Outcome: Day 30 CD3 Donor Chimerism
Description: To measure CD3 donor chimerism post-transplant
Time Frame: 30 days
Measure: Median (Full Range); unit: percentage of chimerism
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
percentage of chimerism | 100 [90 to 100]

5. Secondary Outcome: Day 30 CD33 Donor Chimerism
Description: To measure CD33 donor chimerism at Day 30
Time Frame: 30 days
Measure: Median (Full Range); unit: percentage of chimerism
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
percentage of chimerism | 100 [93 to 100]

6. Secondary Outcome: Graft Versus Host Disease
Description: To measure days to onset of acute graft versus host disease
Time Frame: 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 25
days | 28.5 [22 to 191]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug through 30 days after administration of the last dose of MLN9708.
Description: We used the standard definition of adverse events. Only grade 3-4 adverse events were tracked and reported. Grade 3 & 4 AEs are listed in the 'other non-serious' adverse events as they were documented. They did not meet the definition of serious therefore are listed in the separate category.
Arm/Group | Haploidentical Transplant
All-Cause Mortality (participants affected / at risk) | 8/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant (N=25)
Fever (Infections and infestations) | 10 (15)
Nausea & vomiting (Gastrointestinal disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Graft Versus Host Disease (General disorders) | 2 (2)
DIarrhea (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Bacteremia (Infections and infestations) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
HHV6 infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant (N=25)
Graft versus host disease (General disorders) | 7 (7)
Skin rash with or without pruritis (Skin and subcutaneous tissue disorders) | 8 (8)
Hypertension (Cardiac disorders) | 8 (8)
Elevated AST (Investigations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Hyperglycemia (Investigations) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Syncope (Cardiac disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02169791/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02169791/ICF_001.pdf